CLINICAL TRIAL: NCT05918250
Title: A Phase 1, Open-Label, Multicenter, Study of mRNA-2736 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: mRNA-2736 for Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue development of mRNA-2736 for strategic business reasons.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-2736-P101; 2023-503286-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: mRNA-2736; First-in-human; FIH; Dose-escalation
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-2736 (Experimental): Participants will receive mRNA-2736.
  Interventions: Biological: mRNA-2736

INTERVENTIONS:
Biological: mRNA-2736 — mRNA-2736 will be administered IV.

SUMMARY:
This study is designed to evaluate the safety and tolerability of mRNA-2736 in participants with RRMM.

DETAILED DESCRIPTION:
This open-label, Phase 1, dose-escalation, first-in-human (FIH) clinical study of mRNA-2736 in participants with RRMM is designed to evaluate the safety and tolerability of escalating doses of mRNA-2736, administered intravenously (IV), to determine maximum tolerated dose and/or recommended Phase 2 dose, pharmacokinetics, pharmacodynamics, and preliminary efficacy of mRNA-2736.

ELIGIBILITY:
Key Inclusion Criteria:

* RRMM with prior exposure to a proteasome inhibitor, an immunomodulatory drug (IMiD), and an anti-cluster of differentiation (CD38) monoclonal antibody. Participants must have received at least 3 prior lines of therapy or be triple-class refractory. Participants that are intolerant of a proteasome inhibitor, IMiD, or aCD38 are eligible.
* Measurable disease defined as at least 1 of the following:

  * Serum M-protein ≥0.5 grams/deciliter
  * Urine M-protein ≥200 milligrams (mg)/24 hour
  * Involved free light chain (FLC) ≥100 mg/liter and an abnormal FLC ratio
  * Plasmacytoma with a single diameter ≥2 centimeters
  * Bone marrow plasma cells >30%

Key Exclusion Criteria:

* Known central nervous system (CNS) myeloma or clinical signs and symptoms of CNS involvement of myeloma.
* Active plasma cell leukemia, defined as peripheral blood plasma cells ≥20%. History of plasma cell leukemia is allowed.
* Radiotherapy or cytotoxic chemotherapy within 2 weeks prior to Day 1 (Baseline), except palliative radiotherapy of limited field is permissible within 2 weeks after discussion with the Sponsor medical monitor.
* Antibody-based immunotherapy (monoclonal antibody, bispecific antibody, antibody drug conjugate, radioimmunoconjugate) within 21 days prior to Day 1 (Baseline).
* Proteasome inhibitor therapy within 14 days prior to Day 1 (Baseline).
* Immunomodulatory agent therapy within 7 days of Day 1 (Baseline).
* Autologous hematopoietic cell transplant within 100 days prior to Day 1 (Baseline).
* Allogeneic hematopoietic cell transplant within 180 days prior to Day 1 (Baseline). Participants should have no evidence or ongoing treatment for acute or chronic graft versus host disease.
* Genetically modified adoptive cellular therapy (for example, chimeric antigen receptor T cell, chimeric antigen receptor natural killer) within 12 weeks prior to Day 1 (Baseline).
* Corticosteroid therapy ≥140 mg prednisone or equivalent cumulative dose within 14 days prior to Day 1 (Baseline).
* Active hepatitis B or C, or laboratory evidence for a chronic infection with hepatitis B or C at the time of screening. Participants with a past or resolved hepatitis B infection (presence of hepatitis B core antibody and absence of hepatitis B surface antigen) are eligible. Participants positive for hepatitis C virus (HCV) antibody are eligible only if negative for HCV RNA.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to 1 year

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0 (predose) to 96 hours postdose
Area Under the Concentration-time Curve (AUC) | 0 (predose) to 96 hours postdose
Maximum Effect/Concentration of the Expressed Protein (Emax) | 0 (predose) to 96 hours postdose
Area Under the Effect Concentration (AUEC) | 0 (predose) to 96 hours postdose
Overall Response Rate (ORR) | Up to 2 years
Clinical Benefit Rate (CBR) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Overall Survival (OS) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - UAB Hospital, Birmingham, Alabama
  - University of Miami Health System, Miami, Florida
  - Washington University Medical Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Ohio State University Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - UW Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec